CLINICAL TRIAL: NCT05752708
Title: Evaluation of Perioperative Anxiety Risk Factors in Parents of Children Undergoing Thoracic Surgery
Brief Title: Perioperative Anxiety Risk Factors in Parents of Children Undergoing Thoracic Surgery
Status: Recruiting | Type: Observational
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: KB-74/2022
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-04

CONDITIONS: Anxiety State; Anxiety Postoperative; Parents; Surgery; Thoracic; Satisfaction
Keywords: anxiety, parents, thoracic surgery, perioperative, parents' satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Evaluation of perioperative anxiety in parents of children undergoing thoracic surgery using standardized tests: The Amsterdam Preoperative Anxiety and Information Scale (APAIS), the State-Trait Anxiety Inventory (STAI).

SUMMARY:
Risk factors associated with perioperative anxiety in parents of pediatric patients undergoing thoracic surgery are unknown. It is therefore necessary to identify them in order to better understand, above all, modifiable factors. This will allow the implementation of psychological interventions tailored to the individual needs of parents to strengthen their coping mechanisms before surgery, and thus facilitate the recovery process of their children after surgery.

The purpose of the study is:

1. assessment of the level of anxiety experienced by parents before and after thoracic surgery,
2. assessment of risk factors for parents' perioperative anxiety,
3. assessment of the relationship between parents' perioperative anxiety and satisfaction with postoperative analgesia

DETAILED DESCRIPTION:
According to the literature, parents of children undergoing various types of surgical procedures are accompanied by high levels of anxiety. It was found that the level of anxiety is higher in female parents and is related to the child's age, fear of postoperative pain in children, the scope of information about the course of surgery and anesthesia, and potential complications that may occur during and after the child's operation. Parental anxiety correlates positively with child anxiety. High levels of anxiety in children can lead to many undesirable clinical, psychological and behavioral symptoms during hospitalization (delirium, increased postoperative pain, greater need for analgesia) and after discharge from the hospital (separation anxiety, sleep disorders, aggression, enuresis).

ELIGIBILITY:
Inclusion Criteria:

* parent of child <18 years
* parent of child undergoing thoracic surgery
* parent of child with intravenous or epidural postoperative analgesia
* parent of child with 1-3 score according to the American Society of Anesthesiologists

Exclusion Criteria:

* a parent of a nationality other than Polish
* difficult communication with parent
* parent of a child undergoing oncological treatment
* parent of a child without chest drainage
* lack of parental consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children undergoing thoracic surgery in the Department of Thoracic Surgery of the Institute of Tuberculosis and Lung Disease, Rabka Zdrój Branch.
Sampling Method: Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Parents' anxiety and information requirement in the preoperative phase | before surgery
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) consists of six items. The items are rated on a five point Likert scale with the end poles "not at all" (1) and "extremely" (5). It represents the two scales anxiety (Item 1, 2, 4 and 5) and need-for-information (Items 3 and 6). A total value is calculated by adding up the two scales anxiety and need-for-information. A higher score means higher preoperative anxiety and a greater need for information.
Parents' anxiety state | before surgery, before discharge from the hospital
  Anxiety was determined with a Polish version of the State-Trait Anxiety Inventory (STAI; range: 20-80 pts). The instrument consisting of two separate 20-item scales measuring state and trait anxiety. The results will be expressed as sten scores, from 1-10 (1-4 = low level of anxiety, 5-6 = moderate level of anxiety, >7 = high level of anxiety).

SECONDARY OUTCOMES:
Parents' satisfaction | up to discharge from the hospital
  Satisfaction is assessed on a five-point scale, where 1 means the lowest satisfaction and 5 the highest.
Socio-demographic factors | perioperative period
  Socio-demographic variables include: age, sex, education, marital status, income, place of residence, number of children, number of operations/hospitalizations of the child, scope of information obtained before the operation, postoperative pain and complication in a child

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Tomaszek, PhD, Principal Investigator — National Institute for Tuberculosis and Lung Diseases, Poland
Locations (1):
- National Institute for Tuberculosis and Lung Diseases, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code